CLINICAL TRIAL: NCT05770661
Title: Axial Length Study of Children and Adolescents in Ten Provinces of China
Brief Title: China Axial Length Study
Acronym: CALS
Status: Recruiting | Type: Observational
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Collaborators: Tongji Hospital (Other); Sichuan Provincial People's Hospital (Other); Shandong University of Traditional Chinese Medicine (Other); People's Hospital of Ningxia Hui Autonomous Region (Other); First Affiliated Hospital of Kunming Medical University (Other); The First Affiliated Hospital of Guangxi Traditional Chinese Medical University (Unknown); Affiliated Hospital of Inner Mongolia Minzu University (Unknown); Xinjiang Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Principal Investigator, Jiannan Huang, Doctor, Shanghai Eye Disease Prevention and Treatment Center
Other Study IDs: NO.CALS20220101
Record Dates: First submitted 2023-03-05; First posted 2023-03-15 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Axial Length; Myopia; Child Development
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Myopes: To collect the ocular data among myopic children.
- Non-myopes: To collect the ocular data among non-myopic children.

SUMMARY:
The primary objective of this multi-center, observational study is to establish the reference ranges of axial length in Chinese children and adolescents.

30,000 children aged 3-18 years were examined with cycloplegia to collect their ocular parameters and were all followed up for three years with annual visits.

ELIGIBILITY:
Inclusion Criteria:

* Aged 3 to 18 years
* Have been lived in the research areas for at least one year, and will not move to other places in the following two years
* Parents or guardians sign an informed consent form, and children over 6 years old need oral consent to participate

Exclusion Criteria:

* Mental diseases, unable to cooperate to complete the eye assessment
* Ophthalmic diseases, inability to cooperate to complete the inspection

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Students aged from 3 to 18 years old were recruited from schools to enroll the study.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Axial length | 2023-2026
  Axial length in millimeter was examined by IOL Master

SECONDARY OUTCOMES:
Axial length elongation | 2023-2026
  The elongation in millimeter was the difference between two annual visits.

OTHER OUTCOMES:
Comparison of visual acuity outcomes obtained by VA charts with different optotypes among children | Baseline vision testing at enrollment (single study visit)
  This outcome measure evaluates differences in uncorrected visual acuity (UCVA) results obtained using HOTV and Tumbling E logMAR charts among children aged 3-15 years.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Eye Disease Prevention & Treatment Center, Shanghai, Shanghai Municipality
  - Shanghai Eye Disease Prevention and Treatment Center, Shanghai